CLINICAL TRIAL: NCT06994962
Title: Development and Initial Testing of a Multi-Component Breath Alcohol-Focused Intervention for Young Adults, Stage 3
Brief Title: Multi-Component Breath Alcohol Intervention Phase 3
Acronym: BAMTECH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northeastern University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: IRB24-12-32
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Alcohol Use; Alcohol Drinking; Drinking Behavior
MeSH Terms: conditions — Alcohol Drinking; Drinking Behavior | interventions — Motivational Interviewing; Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Moderate drinking technologies with "lower tech" facilitation (Experimental): Brief motivational-interviewing-based counseling followed by use of three moderate drinking technologies (breath alcohol device and app, blood alcohol content estimator app and self-texting procedure) with "lower tech" facilitation.
  Interventions: Device: Alcohol-related mobile health technologies; Behavioral: Motivational interview and psychoeducation on blood/breath alcohol concentration; Behavioral: Lower tech facilitation
- Moderate drinking technologies with "higher tech" facilitation (Experimental): Brief motivational-interviewing-based counseling followed by use of three moderate drinking technologies (breath alcohol device and app, blood alcohol content estimator app and self-texting procedure) with "higher tech" facilitation
  Interventions: Device: Alcohol-related mobile health technologies; Behavioral: Motivational interview and psychoeducation on blood/breath alcohol concentration; Behavioral: Higher tech facilitation
- Alcohol Education Condition (Active Comparator): Brief session administering non-personalized information about alcohol followed by the option to receive educational alcohol-related information via text
  Interventions: Behavioral: Alcohol Education; Device: Alcohol Education Technology

INTERVENTIONS:
Device: Alcohol-related mobile health technologies — Participants will be asked to use the mobile technologies as they choose while drinking for a four-week period.
  Other Names: Smartphone Breathalyzer; BAC Estimator App; Self-Texting App
  Arms: Moderate drinking technologies with "higher tech" facilitation; Moderate drinking technologies with "lower tech" facilitation
Behavioral: Motivational interview and psychoeducation on blood/breath alcohol concentration — Brief 25/30-minute motivational interview and psychoeducation on blood/breath alcohol concentration that includes both personalized and standardized information.
  Other Names: M.I.
  Arms: Moderate drinking technologies with "higher tech" facilitation; Moderate drinking technologies with "lower tech" facilitation
Behavioral: Lower tech facilitation — Study staff will review instructions for technology use closely with participants and guide them in use of existing phone technologies as reminders for use of the three moderate drinking technologies during drinking situations.
  Arms: Moderate drinking technologies with "lower tech" facilitation
Behavioral: Higher tech facilitation — Participants will use an app developed during the study, SmartSip, that will provide protective behavioral strategies and reminders for use of the three moderate drinking technologies during drinking situations.
  Other Names: SmartSip
  Arms: Moderate drinking technologies with "higher tech" facilitation
Behavioral: Alcohol Education — Brief 25/30-minute psychoeducation on generalized alcohol use providing information about alcohol and its effects, adapted from the National Institute on Alcohol Abuse and Alcoholism (NIAAA) Rethinking Drinking resources
  Arms: Alcohol Education Condition
Device: Alcohol Education Technology — Participants will be able to prompt text messages which will provide them one-off trivia facts using information provided during the attention control psychoeducation session
  Arms: Alcohol Education Condition

SUMMARY:
This is the third stage of a three-stage, NIH-funded study to develop and test a multi-modal intervention concerning blood/breath alcohol concentration for young adults who drink heavily. The multimodal intervention will be made up of brief telehealth counseling and psychoeducation and use of three existing mobile technologies. The brief counseling/psychoeducation and mobile technologies provide personalized feedback regarding blood or breath alcohol content. The long-term goal of use of these mobile technologies will be to facilitate moderate drinking. However, the main goals of the proposed research are to learn more about feasibility of our procedures, perceived value of the technologies and ease of use from the research participants' points of view. In this third stage of the study, the investigators will conduct a randomized controlled trial building on the formative research conducted in Stages 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18-25
* Be able to read English and complete study evaluations
* At least occasional heavy episodic drinking (i.e., 4 or more drinks for women and 5 or more drinks for men) over the prior 30 days
* Frequent consumption of at least one alcoholic drink during a minimum of 12 days out of the prior 30 so that subjects will have multiple opportunities to use the moderate drinking technologies during the intervention period.

Exclusion Criteria:

* Severe substance use disorder
* Be psychotic or otherwise severely psychiatrically disabled
* Report a history of a medical condition that would contraindicate the consumption of alcohol (e.g., liver disease, cardiac abnormality, pancreatitis, diabetes, neurological problems, and gastrointestinal disorders)

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Technology utilization | 4-week field use period
  Percentage of reported drinking days on which one reports that moderate drinking technology use has occurred
Acceptability | 4-week field use period
  Score on acceptability subscale of Modified System Usability Scale
Usability | 4-week field use period
  Score on acceptability subscale of Modified System Usability Scale

SECONDARY OUTCOMES:
Drinks per drinking day | 4-week field use period
  Number of drinks per day during field testing period
Estimated blood alcohol content | 4-week field use period
  Average estimated blood alcohol content reached on drinking days
Negative Consequences | 4-week field use period
  Score on the Young Adult Alcohol Consequences Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Robert F Leeman, Ph.D., Principal Investigator — Northeastern University
Locations (1):
- Northeastern University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Study materials and datasets with identifiers removed will be shared with other investigators upon request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Study materials are available to qualified investigators at any time upon request. Datasets with identifiers removed will be available after publication of the main outcome paper from the study
Access Criteria: Any qualified investigator upon request